CLINICAL TRIAL: NCT02763852
Title: Pharmacokinetic-Pharmacodynamic Interaction Between Four Different Single Doses of BIA 3-202 and a Single Dose of Levodopa/Benserazide (100/25 mg): a Double-blind, Randomised, Crossover, Placebo Controlled Study in Healthy Volunteers
Brief Title: Pharmacokinetic-Pharmacodynamic Interaction Between Four Different Single Doses of BIA 3-202 and a Single Dose of Levodopa/Benserazide (100/25 mg)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bial - Portela C S.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: BIA-3202-104
Record Dates: First submitted 2016-05-04; First posted 2016-05-05 (Estimated); Last update posted 2016-05-05 (Estimated); Status verified 2016-05

CONDITIONS: Parkinson's Disease
Keywords: Parkinson's Disease; Nebicapone
MeSH Terms: conditions — Parkinson Disease | interventions — nebicapone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (5):
- BIA 3-202 50 mg (Experimental): BIA 3-202 single-dose plus 1 tablet of Madopar 125. BIA 3-202 50 mg: 5 tablets of 10 mg. The investigational products were administered orally, following an overnight fast of at least 7 hours, with approximately 200 mL of potable water.
  Interventions: Drug: BIA 3-202; Drug: Madopar® 125
- BIA 3-202 100 mg (Experimental): BIA 3-202/Placebo single-dose plus 1 tablet of Madopar 125. BIA 3-202 100 mg: 1 tablet of 100 mg + 4 placebo tablets. The investigational products were administered orally, following an overnight fast of at least 7 hours, with approximately 200 mL of potable water.
  Interventions: Drug: BIA 3-202; Drug: Placebo; Drug: Madopar® 125
- BIA 3-202 200 mg (Experimental): BIA 3-202/Placebo single-dose plus 1 tablet of Madopar 125. BIA 3-202 200 mg: 2 tablet of 100 mg + 3 placebo tablets. The investigational products were administered orally, following an overnight fast of at least 7 hours, with approximately 200 mL of potable water
  Interventions: Drug: BIA 3-202; Drug: Placebo; Drug: Madopar® 125
- BIA 3-202 300 mg (Experimental): BIA 3-202/Placebo single-dose plus 1 tablet of Madopar 125. BIA 3-202 300 mg: 3 tablet of 100 mg + 2 placebo tablets. The investigational products were administered orally, following an overnight fast of at least 7 hours, with approximately 200 mL of potable water.
  Interventions: Drug: BIA 3-202; Drug: Placebo; Drug: Madopar® 125
- BIA 3-202 400 mg (Experimental): BIA 3-202/Placebo single-dose plus 1 tablet of Madopar 125. BIA 3-202 400 mg: 4 tablet of 100 mg + 1 placebo tablets. The investigational products were administered orally, following an overnight fast of at least 7 hours, with approximately 200 mL of potable water
  Interventions: Drug: BIA 3-202; Drug: Placebo; Drug: Madopar® 125

INTERVENTIONS:
Drug: BIA 3-202 — The study consisted of 5 treatment periods. Eligible subjects were admitted to the UFH on the morning of the day prior to receive the trial medication (dosing day) and remained in the unit for at least 30 h post-dose.
  Subjects were to receive BIA 3-202 50 mg, 100 mg, 200 mg, 400 mg and placebo at 5 separate treatment periods.
Drug: Placebo — Placebo dose consisted of 5 tablets matching BIA 3-202 100 mg tablets; oral route.
  Arms: BIA 3-202 100 mg; BIA 3-202 200 mg; BIA 3-202 300 mg; BIA 3-202 400 mg
Drug: Madopar® 125 — Levodopa 100 mg/benserazide 25 mg capsules (Madopar® 125, marketed by Roche products Limited); oral route.

SUMMARY:
The purpose of this study is to investigate the tolerability, pharmacokinetic profile of BIA 3-202 and its metabolites, and the pharmacokinetic and pharmacodynamic interaction between 4 different single doses of BIA 3-202 (50 mg, 100 mg, 200 mg and 400 mg) and a single dose of standard levodopa 100 mg/benserazide 25 mg (Madopar® 125) in adult male and female healthy volunteers.

DETAILED DESCRIPTION:
This was a single centre, double-blind, randomised, placebo-controlled, single-graded-dose, crossover study with five single-dose treatment periods. The washout period between doses was 15±2 days. For each of the five treatment periods, volunteers were to be admitted at the UFH on the day before the treatment day. On each treatment period, the pre-dose assessment were to be completed, BIA 3-202/Placebo was to be administered concomitantly with the dose of Madopar® 125 and post-dose assessments were to be completed. Subjects were discharged 30 h post-dose. Subjects should attend five treatment periods and were to receive a different dose of BIA 3-202 or placebo during each of these treatment periods.

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects aged between 18 and 45 years, inclusive.
* Subjects of body mass index (BMI) between 19 and 28 kg/m2, inclusive.
* Subjects who were healthy as determined by pre study medical history, physical examination, and 12- lead ECG.
* Subjects who had clinical laboratory tests acceptable to the investigator.
* Subjects who were negative for HBsAg, anti-HCV Ab and HIV-1 and HIV-2 Ab tests at screening.
* Subjects who were negative for drugs of abuse at screening and admission.
* Subjects who were non-smokers or who smoked less than 10 cigarettes or equivalent per day.
* Subjects who were able and willing to give written informed consent.
* (If a woman) She was not of childbearing potential by reason of surgery or, if of childbearing potential, she used one of the following methods of contraception: double barrier, intrauterine device or abstinence.

Exclusion Criteria:

Subjects who did not conform to the above inclusion criteria, OR

* Subjects who had a clinically relevant history or presence of respiratory, gastrointestinal, renal, hepatic, haematological, lymphatic, neurological, cardiovascular, psychiatric, musculoskeletal, genitourinary, immunological, dermatological, connective tissue diseases or disorders.
* Subjects who had a clinically relevant surgical history.
* Subjects who had a clinically relevant family history.
* Subjects who had a history of relevant atopy.
* Subjects who had a history of relevant drug hypersensitivity.
* Subjects who had a history of alcoholism or drug abuse.
* Subjects who consumed more than 28 units of alcohol a week.
* Subjects who had a significant infection or known inflammatory process on screening and/or admission.
* Subjects who had acute gastrointestinal symptoms at the time of screening and/or admission (e.g., nausea, vomiting, diarrhoea, heartburn).
* Subjects who had an acute infection such as influenza at the time of screening and/or admission.
* Subjects who had used prescription drugs within 4 weeks of first dosing.
* Subjects who had used oral contraceptives or over the counter medication excluding oral routine vitamins but including mega dose vitamin therapy within one week of first dosing.
* Subjects who had used any investigational drug and/or participated in any clinical trial within 3 months of their first admission to the study.
* Subjects who had previously received BIA 3-202.
* Subjects who had donated and/or received any blood or blood products within the previous 3 months prior to screening.
* Subjects who were vegetarians, vegans and/or had medical dietary restrictions.
* Subjects who could not communicate reliably with the investigator.
* Subjects who were unlikely to co-operate with the requirements of the study.
* (If woman) She was pregnant or breast-feeding.
* (If woman) She was at childbearing potential and she did not use an approved effective contraceptive method or she used oral contraceptives.
* Subjects who were unwilling or unable to give written informed consent.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2001-04; Primary Completion 2001-07 (Actual); Study Completion 2001-07 (Actual)

PRIMARY OUTCOMES:
Maximum observed plasma concentration (Cmax) | pre-dose, ½, 1, 1½, 2, 3, 4, 6, 8, 12, 18 and 24 h post-dose
Area under the plasma concentration time curve extrapolated to infinity (AUC0-∞) | pre-dose, ½, 1, 1½, 2, 3, 4, 6, 8, 12, 18 and 24 h post-dose
Apparent terminal elimination half-life (t1/2) | pre-dose, ½, 1, 1½, 2, 3, 4, 6, 8, 12, 18 and 24 h post-dose

CONTACTS AND LOCATIONS:
Locations (1):
- Human Pharmacology Unit - BIAL - Portela & Ca, S.A., S. Mamede Do Coronado, S. Mamede Do Coronado, Portugal

IPD SHARING:
Plan to Share IPD: No